CLINICAL TRIAL: NCT01985659
Title: Cohort Analysis of Nodal Upstaging in the Era of Increase of VATS Anatomical Resections for NSCLC
Brief Title: Nodal Upstaging in VATS Anatomical Resections for NSCLC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Principal Investigator, Johnny Moons, RN, MScN, University Hospital, Gasthuisberg
Other Study IDs: pN+VATS
Record Dates: First submitted 2013-11-10; First posted 2013-11-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Lymph Node Excision; Thoracic Surgical Procedures; Thoracic Surgery, Video-Assisted; Thoracotomy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- open thoracotomy: In the first cohort(20007-2009) almost all patients where operated through a thoracotomy.
- Early VATS: In a second cohort, (2010-2011) the experience with vats was early.
- Standardized VATS: In the third period (2012-2013), a standardized vats technique with extensive intrapulmonary and mediastinal lymphadenectomy was used.

SUMMARY:
This study investigates peropeative nodal upstaging during anatomical resections for non-small-cell-lung-cancer in an era of rising numbers of VATS anatomical resections. In case of comparable study groups, unchanged pretreatment staging and equal quality of pathologic examination, lymph node upstaging is a marker of surgical quality and can be used to study the quality of a new surgical technique.

DETAILED DESCRIPTION:
Vats lobectomy is becoming the standard of care for early stage lung cancer. Several studies have shown feasibility and safety in dedicated centres. Compared to thoracotomy the procedure is believed to achieve equal oncologic results and survival, perhaps better.

Publications have shown that mediastianal lymph node dissection during VATS is similar.

However, two recent reports have shown potential lower N1 (hilar and intrapulmonary) upstaging in VATS surgery After optimal staging the percentage of unforeseen N+ the percentage of unforeseen positive nodes can reach 15%

Nodal upstaging at final pathology is dependent on the quality of:

* pretreatment staging, the better, the less upstaging
* surgery, ie mediastinal, hilar and intrapulmonary lymphadenectomy
* pathologic examination If we accept that pretreatment staging and pathologic examination are equal in two comparable surgical cohorts, the finding of unforeseen N+ or nodal upstaging is a quality marker of surgery. When surgical techniques are changing, it is important to look at this marker.

In absence of a randomized trial, we believe a cohort analysis is useful. By including all patients, open or vats, and comparing cohorts instead of the surgical technique used, the selection bias is absent. We compare three cohorts. In the first (20007-2009) almost all patients where operated through a thoracotomy. In a second cohort, (2010-2011) the experience with vats was early. In the third period (2012-2013), a standardized vats technique with extensive intrapulmonary and mediastinal lymphadenectomy was used.

ELIGIBILITY:
Inclusion Criteria:

* All cN0, cN1 patients that underwent segmentectomy, lobectomy, sleeve lobectomy for NSCLC.

Exclusion Criteria:

* cN2
* cM+
* Pneumonectomy
* Previous lung cancer surgery - lymphadenectomy
* Neo-adjunvant therapy
* Lung Tx
* Bilateral lesions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: By including all patients, open or VATS, and comparing cohorts instead of the surgical technique used, the selection bias is absent. We compare three cohorts. In the first (20007-2009) almost all patients where operated through a thoracotomy. In a second cohort, (2010-2011) the experience with vats was early. In the third period (2012-2013), a standardized vats technique with extensive intrapulmonary and mediastinal lymphadenectomy was used.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2013-11; Primary Completion 2014-02 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
proportion of N upstaging | at time of surgical resection
  clinical N0 to pathological N1 clinical N0 to pathological N2 clinical N1 to pathological N2

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Decaluwé, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Alessia Stanzi, MD, Principal Investigator — Universitaire Ziekenhuizen KU Leuven; Christophe Dooms, MD, PhD, Study Chair — Universitaire Ziekenhuizen KU Leuven; Paul De Leyn, MD, PhD, Study Director — Universitaire Ziekenhuizen KU Leuven
Locations (1):
- University Hospital Leuven, Leuven, Belgium